CLINICAL TRIAL: NCT03449979
Title: Rational Optimization of tACS for Targeting Thalamo-Cortical Oscillations (Experiment 3)
Brief Title: Single Session of tACS in a Depressive Episode
Acronym: SSDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16-1911b; R01MH101547 (NIH)
Record Dates: First submitted 2018-02-15; First posted 2018-02-28 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2019-09

CONDITIONS: Depression; Major Depressive Disorder; Premenstrual Dysphoric Disorder; Depressive Episode
Keywords: tACS; transcranial alternating current stimulation; stimulation; heart rate variability; electroencephalogram; EEG
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Premenstrual Dysphoric Disorder

STUDY DESIGN:
Intervention Model Description: This study recruits both participants currently experiencing a depressive episode (regardless of diagnosis) and those with no history of neurological or psychiatric illness. Randomization will occur in a 1:1 ratio for both of these groups, with half of each group receiving transcranial alternating current stimulation (tACS) at 10 Hz and the other half receiving placebo (or sham) stimulation.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study, meaning that neither the participant nor the experimenter knows what kind of stimulation the participant is receiving. An unblinded monitor (separate from the staff that interacts with the participant) is responsible for creating the stimulation codes that run each session and for ensuring that these codes worked correctly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- alpha stimulation in participants in a depressive episode (Experimental): Participants in a depressive episode will receive 2 mA of alternating current stimulation at individualized alpha stimulation (between 8 and 12Hz; determined by an EEG recording prior to stimulation) for 40 minutes. tACS stimulation is delivered using the XCSITE100 Stimulator tACS.
  Interventions: Device: XCSITE100 Stimulator tACS
- sham stimulation in participants in a depressive episode (Placebo Comparator): Sham Stimulation mimics the physical effects of stimulation, with up to one minute of stimulation during the session. Sham stimulation to participants in a depressive episode is delivered using the XCSITE100 Stimulator Sham.
  Interventions: Device: XCSITE100 Stimulator Sham
- alpha stimulation in healthy participants (Experimental): Healthy participants will receive 2 mA of alternating current stimulation at individualized alpha stimulation (between 8 and 12Hz; determined by an EEG recording prior to stimulation) for 40 minutes. tACS stimulation is delivered using the XCSITE100 Stimulator tACS.
  Interventions: Device: XCSITE100 Stimulator tACS
- sham stimulation in healthy participants (Placebo Comparator): Sham Stimulation mimics the physical effects of stimulation, with up to one minute of stimulation during the session. Sham stimulation to healthy participants is delivered using the XCSITE100 Stimulator Sham.
  Interventions: Device: XCSITE100 Stimulator Sham

INTERVENTIONS:
Device: XCSITE100 Stimulator Sham — The participant will receive up to one minute of tACS stimulation until the stimulation fades. Sham stimulation mimics the skin sensations a participant would experience during a tACS session.
  Other Names: Sham tACS
  Arms: sham stimulation in healthy participants; sham stimulation in participants in a depressive episode
Device: XCSITE100 Stimulator tACS — Transcranial alternating current stimulation (tACS) is a method of noninvasive brain stimulation in which weak electrical current are applied to the scalp in a sine wave pattern to induce cortical oscillations at the frequency at which they are applied.
  Other Names: tACS
  Arms: alpha stimulation in healthy participants; alpha stimulation in participants in a depressive episode

SUMMARY:
Purpose: Investigating the effects of non-invasive transcranial alternating current stimulation (tACS) on healthy participants and participants with mood disorders.

Participants: 40 males and females, ages 18-65, with depressed mood; 40 healthy males and females, ages 18-65, free of neurological or psychiatric conditions.

Procedures: This is a single visit study with two stimulation conditions (tACS and sham tACS). The session will begin with clinical assessments (including confirmation of diagnosis), followed by an interactive EEG task, then a 7 minute resting state EEG (2 minutes eyes closed, 5 minutes eyes open), followed by the stimulation session (40 minutes of tACS or sham tACS), followed by an additional 5 minute resting state EEG. The stimulation will involved 40 minutes of transcranial alternating current stimulation, 2 mA in amplitude and at individualized alpha frequency (determined by the 2 minutes eyes closed EEG recording; between 8 and 12Hz).

DETAILED DESCRIPTION:
Participants will report for a study visit and will review and sign a consent form.

Participants will complete several clinical assessments and also take a urine drug test and urine pregnancy test (if applicable). Eligibility will be re-assessed by the investigators before the participant moves on to the next phase.

If the participant still qualifies, the participant will first be fitted with two 5x5cm electrodes placed over F3/F4 (10-20 measurement system) and one 5x7cm electrode placed over Cz. In addition, the participant will have a 128-channel EEG net placed on their head. Participants will provide a saliva sample to assess for brain-derived neurotrophic factor (BDNF), which may affect how the participant's brain responds to stimulation. Once the participant is fitted with this equipment, the participant will complete two interactive EEG tasks, then 2-minute resting state EEG with the participant's eyes closed, then a 5-minute resting state EEG with the participant's eyes open.

Following these recordings, participants will respond to additional questionnaires. Immediately following this, the participant will receive 40 minutes of stimulation (tACS or sham tACS). During this stimulation, participants will sit comfortably upright and awake.

After stimulation has completed, participants will respond to additional questionnaires. Once completed, participants will then complete an additional 5-minute resting state EEG with the participant's eyes open, as well as complete one of the additional interactive EEG tasks.

Finally, participants will respond to a blinding questionnaire to assess if the participant thought that the participant received stimulation. Once complete, the participant will leave. This session is estimated to last about 4 hours.

ELIGIBILITY:
Inclusion Criteria for individuals with depressed mood:

* Ages 18-65 years
* Hamilton Depression Rating Scale score >8
* Capacity to understand all relevant risks and potential benefits of the study (informed consent)
* Low suicide risk which will be determined through the use of both the Structured Clinical Interview for the DSM-5 and by scoring less than 3 (0,1, or 2) in the Hamilton rating depression scale.
* Negative pregnancy test for female participants

Exclusion Criteria for individuals with depressed mood:

* DSM-5 diagnosis of alcohol of substance abuse (other than nicotine) within the 12 months
* DSM-5 diagnosis of alcohol or substance dependence (other than nicotine) within the last 12 months
* DSM-5 diagnosis of personality disorder
* Eating disorder (current or within the past 3 months)
* Anything that, in the opinion of the investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the study
* Neurological disorders, including but not limited to history of seizures (except childhood febrile seizures and electro-convulsive therapy (ECT) induced seizures), dementia, history of stroke, Parkinson's disease, multiple sclerosis, cerebral aneurysm.
* Medical or neurological illness (unstable cardiac disease, AIDS, malignancy, liver or renal impairment) or treatment for a medical disorder that could interfere with study participation
* History of traumatic brain injury, reoccurring seizures or later cognitive rehabilitation or causing cognitive sequelae
* History of childhood trauma (determined by the Childhood Trauma Questionnaire)
* Prior brain surgery
* Any brain devices/implants, including cochlear implants and aneurysm clips
* Co-morbid neurological condition (i.e. seizure disorder, brain tumor)
* Use of illicit drugs, confirmed by a drug test
* Non English speakers
* Pregnant or nursing females
* Current use of benzodiazepines or anti-epileptic drugs

Inclusion Criteria for healthy controls:

* Ages 18-65 years
* Hamilton Depression Rating Scale score ≤8
* Capacity to understand all relevant risks and potential benefits of the study (informed consent)
* Negative pregnancy test for female participants

Exclusion Criteria for healthy controls:

* History of major neurological or psychiatric illness, including epilepsy
* Medication use associated with neurological or psychiatric illnesses
* Currently undergoing counseling or psychotherapy treatment for depression, anxiety, eating disorders, PTSD or other behavioral conditions
* DSM-5 diagnosis of personality disorder
* First degree relative (parent, sibling, child) with major neurological or psychiatric illness
* Prior brain surgery
* Major head injury
* Any brain devices/implants (including cochlear implants and aneurysm clips)
* History of childhood trauma (determined by the Childhood Trauma Questionnaire)
* Use of illicit drugs, confirmed by a drug test
* Braids or other hair styling that prevents direct access to the scalp (if removal not possible)
* Skin allergies or very sensitive skin
* Non English speakers
* Pregnant or nursing females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Alpha Stimulation in Participants in a Depressive Episode: Participants in a depressive episode will receive 2 mA of alternating current stimulation at individualized alpha stimulation (between 8 and 12 Hz; determined by an EEG recording prior to stimulation) for 40 minutes. tACS stimulation is delivered using the XCSITE100 Stimulator tACS.
  XCSITE100 Stimulator tACS: Transcranial alternating current stimulation (tACS) is a method of noninvasive brain stimulation in which weak electrical current are applied to the scalp in a sine wave pattern to induce cortical oscillations at the frequency at which they are applied.
- Alpha Stimulation in Healthy Participants: Healthy participants will receive 2 mA of alternating current stimulation at individualized alpha stimulation (between 8 and 12 Hz; determined by an EEG recording prior to stimulation) for 40 minutes. tACS stimulation is delivered using the XCSITE100 Stimulator tACS.
  XCSITE100 Stimulator tACS: Transcranial alternating current stimulation (tACS) is a method of noninvasive brain stimulation in which weak electrical current are applied to the scalp in a sine wave pattern to induce cortical oscillations at the frequency at which they are applied.
Period: Overall Study
Arm/Group | Alpha Stimulation in Participants in a Depressive Episode | Sham Stimulation in Participants in a Depressive Episode | Alpha Stimulation in Healthy Participants | Sham Stimulation in Healthy Participants
Started | 21 | 20 | 21 | 22
Completed | 21 | 20 | 21 | 21
Not Completed | 0 | 0 | 0 | 1
Not completed — Technical difficulty | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: One healthy control participant that received sham stimulation was excluded from analysis as we were unable to find an age and sex matched participant. One healthy control participant that received sham stimulation did not complete the study due to technical difficulties.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alpha Stimulation in Participants in a Depressive Episode | Sham Stimulation in Participants in a Depressive Episode | Alpha Stimulation in Healthy Participants | Sham Stimulation in Healthy Participants | Total
Number analyzed (Participants) | 21 | 20 | 21 | 22 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.429 (11.902) | 27.65 (12.227) | 28.095 (11.432) | 27.182 (12.133) | 27.796 (11.831)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 17 | 17 | 67
  Male | 4 | 4 | 4 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 6 | 2 | 9
  Not Hispanic or Latino | 20 | 19 | 14 | 17 | 70
  Unknown or Not Reported | 1 | 0 | 1 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 4 | 7 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 2 | 4 | 12
  White | 15 | 16 | 13 | 10 | 54
  More than one race | 1 | 1 | 2 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 20 | 21 | 22 | 84
Alpha oscillations in left frontal cortex before stimulation [Mean (Standard Deviation); unit: microvolts] — Population: One healthy control participant that received sham stimulation was excluded from analysis as we were unable to find an age and sex matched participant. One healthy control participant that received sham stimulation did not complete the study due to technical difficulties.
  microvolts
    number analyzed (Participants) | 21 | 20 | 21 | 20 | 82
    (all) | 0.789 (0.088) | 0.812 (0.056) | 0.826 (0.076) | 0.845 (0.095) | 0.818 (0.081)

OUTCOME MEASURES:

1. Primary Outcome: Change in Alpha Frequency Electrical Activity in Left Frontal Cortex From Stimulation
Description: Fast Fourier transform is applied to 5 minutes of EEG data before and after intervention. Primary outcome is the difference in alpha frequency amplitude (8-12 Hz) in the left frontal cortex from baseline as a result of intervention.
Time Frame: 5 minute recording before and after intervention
Population: One of the healthy participants that received sham stimulation could not be age and sex matched, therefore, we did not analyze this participant.
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Alpha Stimulation in Participants in a Depressive Episode | Sham Stimulation in Participants in a Depressive Episode | Alpha Stimulation in Healthy Participants | Sham Stimulation in Healthy Participants
Number analyzed (Participants) | 21 | 20 | 21 | 20
microvolts | -0.005 (0.022) | 0.008 (0.023) | 0.004 (0.017) | 0.007 (0.022)
Statistical Analysis 1: Comparison: Alpha Stimulation in Participants in a Depressive Episode vs Sham Stimulation in Participants in a Depressive Episode; Interaction in the effect of tACS on left frontal alpha oscillation in the depressed group. Two-way interaction of within-participant factor of before/after tACS and between-participant factor of alpha-tACS/placebo; Test type: Superiority; p = 0.0852, ANOVA; degrees of freedom = (1,39); F-statistic = 3.119
Statistical Analysis 2: Comparison: Alpha Stimulation in Healthy Participants vs Sham Stimulation in Healthy Participants; Interaction in the effect of tACS on left frontal alpha oscillation in the healthy group. Two-way interaction of within-participant factor of before/after tACS and between-participant factor of alpha-tACS/placebo; Test type: Superiority; p = 0.6676, ANOVA; degrees of freedom = (1,39); F-statistic = 0.187
Statistical Analysis 3: Comparison: Alpha Stimulation in Participants in a Depressive Episode vs Alpha Stimulation in Healthy Participants; Main effect of alpha-tACS on session (before and after) on left frontal alpha oscillations across both groups (healthy and patient); Test type: Superiority; p = 0.929, ANOVA — degrees of freedom = (1,41); F-statistic = 0.008
Statistical Analysis 4: Comparison: Alpha Stimulation in Participants in a Depressive Episode; Difference in alpha oscillations after versus before in the depressed cohort (one-tailed Student's t-test) with the hypothesis to decrease pathologically elevate left frontal alpha oscillations; Test type: Superiority; p = 0.1950, t-test, 1 sided; degrees of freedom = 20; t-statistic = -0.08789
Statistical Analysis 5: Comparison: Alpha Stimulation in Healthy Participants; Difference in alpha oscillations after versus before in the healthy cohort (one-tailed Student's t-test) run as a control analysis; Test type: Superiority; p = 0.8603, t-test, 1 sided; degrees of freedom = 20; t-statistic = 1.1117

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 5 hours of the single session experiment
Groups:
- Alpha Stimulation in Patients in a Depressive Episode: Participants in a depressive episode will receive 2 mA of alternating current stimulation at individualized alpha stimulation (between 8 and 12 Hz; determined by an EEG recording prior to stimulation) for 40 minutes. tACS stimulation is delivered using the XCSITE100 Stimulator tACS.
  XCSITE100 Stimulator tACS: Transcranial alternating current stimulation (tACS) is a method of noninvasive brain stimulation in which weak electrical current are applied to the scalp in a sine wave pattern to induce cortical oscillations at the frequency at which they are applied.
- Sham Stimulation in Patients in a Depressive Episode: Sham Stimulation mimics the physical effects of stimulation, with up to one minute of stimulation during the session. Sham stimulation to participants in a depressive episode is delivered using the XCSITE100 Stimulator Sham.
  XCSITE100 Stimulator Sham: The participant will receive up to one minute of tACS stimulation until the stimulation fades. Sham stimulation mimics the skin sensations a participant would experience during a tACS session.
Arm/Group | Alpha Stimulation in Patients in a Depressive Episode | Sham Stimulation in Patients in a Depressive Episode | Alpha Stimulation in Healthy Participants | Sham Stimulation in Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 12/21 | 7/20 | 9/21 | 5/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha Stimulation in Patients in a Depressive Episode (N=21) | Sham Stimulation in Patients in a Depressive Episode (N=20) | Alpha Stimulation in Healthy Participants (N=21) | Sham Stimulation in Healthy Participants (N=22)
Tingling (Investigations) | 7 (7) | 2 (2) | 7 (7) | 4 (4)
Flickering Lights (Investigations) | 3 (3) | 0 (0) | 3 (3) | 2 (2)
Itching (Investigations) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Burning sensation (Investigations) | 7 (7) | 3 (3) | 3 (3) | 3 (3)
Scalp pain (Investigations) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Neck pain (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/79/NCT03449979/Prot_SAP_000.pdf